CLINICAL TRIAL: NCT00858858
Title: Clinical Studies on Bile Acids in Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GAST-002-08F; NCT00849420 (obsolete NCT alias)
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): All patients are treated with DCA and UDCA perfusion of the esophagus, one year apart, followed by 8 weeks of treatment with oral ursodeoxycholic acid 10 mg/kg qd. Then a final DCA perfusion of the esophagus.
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — 8 weeks of oral UDCA treatment 10 mg/kg qd
  Other Names: UDCA

SUMMARY:
This study has two major goals:

1. To determine the effects of bile salts on causing DNA injury and activating signaling pathways that promote growth in cells from the esophagus of patients who have gastroesophageal reflux disease (GERD)
2. To determine whether changes in bile composition induced by treating patients with a bile salt called ursodeoxycholic acid (UDCA) can alter DNA injury, signaling pathway activation and other types of damage in cells from the esophagus of patients who have GERD.

DETAILED DESCRIPTION:
Patients who have been scheduled for elective endoscopic examination at the Dallas VA Medical Center for the evaluation of GERD or Barrett's esophagus will be invited to participate in the study. Patients who provide written, informed consent will have a medical history taken.

Women of child bearing potential will have a pregnancy test. Eligible subjects will be treated with omeprazole 20 mg BID for at least four weeks before the scheduled endoscopic examination. Eight days before the endoscopy, patients will be instructed to discontinue any aspirin and other non-steroidal anti-inflammatory drugs (unless there is a contraindication to discontinuing those medications including a history of coronary artery disease, myocardial infarction, cerebrovascular accident or transient ischemic attacks). The endoscopic examination, which had been scheduled for clinical purposes, will be performed as usual, with biopsy specimens taken as required for clinical purposes.

When the clinical examination has been completed, a perfusion catheter will be passed through the biopsy channel and positioned 5 cm above the squamocolumnar junction in the distal esophagus. The distal esophagus will be perfused with 10cc of a 250 M solution of either deoxycholic acid (DCA) or ursodeoxycholic acid (UDCA) for 5 minutes. Odd-number patients enrolled in each of the two patient groups (GERD patients with and without Barrett's esophagus) will receive DCA, whereas even-number patients will receive UDCA. The catheter position, bile acid concentration and duration of bile acid perfusion are chosen to simulate a typical episode of gastroesophageal reflux.

In all patients, 12 biopsy specimens of the squamous epithelium will be taken using jumbo biopsy forceps at a level 2 cm proximal to the squamocolumnar junction at baseline (6 biopsies will be used to establish the primary cell cultures and six will be used for the molecular analyses); 6 more biopsy specimens will be taken at the same level immediately after bile acid perfusion for molecular analyses.

In the patients with Barrett's esophagus, 12 biopsy specimens of the specialized intestinal metaplasia also will be taken using jumbo biopsy forceps at a level 1 cm distal to the squamocolumnar junction at baseline (6 biopsies will be used to establish the primary cell cultures and six will be used for the molecular analyses); 6 more biopsy specimens will be taken a t the same level immediately after bile acid perfusion for molecular analyses. All endoscopic procedures will be performed by Dr. S.J. Spechler.

All patients will be maintained on omeprazole 20 mg BID for one year, after which the endoscopic examinations will be repeated. The endoscopies will be performed with bile acid perfusions and biopsy sampling exactly as described above, except that patients who received DCA during the first examination will receive UDCA and vice-versa.

After the second endoscopy, patients will be treated with UDCA in a dose of 10 mg/kg for 8 weeks, after which a final endoscopy will be performed.

During this endoscopy, DCA perfusion will be performed as described above. In all patients, 6 biopsy specimens of the squamous epithelium will be taken using jumbo biopsy forceps at a level 2 cm proximal to the squamocolumnar junction at baseline for the molecular analyses; 6 more biopsy specimens will be taken at the same level immediately after bile acid perfusion for molecular analyses.

In the patients with Barrett's esophagus, 6 biopsy specimens of the specialized intestinal metaplasia also will be taken using jumbo biopsy forceps at a level 1 cm distal to the squamocolumnar junction at baseline for the molecular analyses; 6 more biopsy specimens will be taken at the same level immediately after bile acid perfusion for molecular analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been scheduled for elective endoscopic examination at the Dallas VA Medical Center for the evaluation of GERD or Barrett's esophagus

Exclusion Criteria:

* Patients unwilling or unable to provide informed consent
* Patients with esophageal carcinomas
* Patients with esophageal varices
* Patients taking warfarin or clopidogrel
* Coagulopathy that precludes safe biopsy of the esophagus
* Comorbidity that precludes safe participation in the study
* Allergy to omeprazole or UDCA
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Spechler, MD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (1):
- VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas, United States

REFERENCES:
- [Background] Huo X, Juergens S, Zhang X, Rezaei D, Yu C, Strauch ED, Wang JY, Cheng E, Meyer F, Wang DH, Zhang Q, Spechler SJ, Souza RF. Deoxycholic acid causes DNA damage while inducing apoptotic resistance through NF-kappaB activation in benign Barrett's epithelial cells. Am J Physiol Gastrointest Liver Physiol. 2011 Aug;301(2):G278-86. doi: 10.1152/ajpgi.00092.2011. Epub 2011 Jun 2. PMID 21636532
- [Derived] Peng S, Huo X, Rezaei D, Zhang Q, Zhang X, Yu C, Asanuma K, Cheng E, Pham TH, Wang DH, Chen M, Souza RF, Spechler SJ. In Barrett's esophagus patients and Barrett's cell lines, ursodeoxycholic acid increases antioxidant expression and prevents DNA damage by bile acids. Am J Physiol Gastrointest Liver Physiol. 2014 Jul 15;307(2):G129-39. doi: 10.1152/ajpgi.00085.2014. Epub 2014 May 22. PMID 24852569

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Esophageal biopsy: After the esophageal perfusions described above, 12 biopsy specimens of the squamous epithelium will be taken at a level 2 cm proximal to the squamocolumnar junction at baseline (6 biopsies will be used to establish primary cell cultures and six will be used for molecular analyses); 6 more biopsy specimens will be taken at the same level immediately after bile acid perfusion for molecular analyses. In patients with Barrett's esophagus, 12 biopsy specimens of the specialized intestinal metaplasia also will be taken at a level 1 cm distal to the squamocolumnar junction at baseline (6 biopsies will be used to establish primary cell cultures and six will be used for molecular analyses); 6 more biopsy specimens will be taken at the same level immediately after bile acid perfusion for molecular analyses.
Period: Overall Study
Arm/Group | Arm 1
Started | 60
Completed | 42
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Protection Against DNA Damage by UDCA
Description: p-H2AX levels are a measure of DNA damage. Our major outcome measure is the change in p-H2AX levels, expressed as relative densitometry units, after DCA perfusion in patients treated with oral UDCA. If UDCA protects against bile acid-induced DNA damage, then p-H2AX levels before and after perfusion should not change significantly.
Time Frame: After 8 weeks of UDCA treatment
Population: Patients with Barrett's esophagus, only metaplastic epithelium evaluated. No data were collected from squamous epithelium as originally planned because our in vitro studies subsequently showed that DCA exposure did not cause DNA damage in squamous cells and, therefore, oral UDCA treatment would be meaningless for squamous esophagus.
Measure: Mean (Standard Error); unit: Relative Densitometry Units
Arm/Group | Arm 1
Number analyzed (Participants) | 21
Relative Densitometry Units
  Before DCA Perfusion | 1.068 (.17)
  After DCA Perfusion | .82 (.14)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=42)
Ruptured cerebral aneurysm (Vascular disorders) | 1 (1) — SAE unrelated to study intervention.
Ischemic colitis (Gastrointestinal disorders) | 1 (1) — SAE unrelated to study intervention
Death (Cardiac disorders) | 1 (1) — SAE unrelated to study intervention
Abdominal pain (Gastrointestinal disorders) | 1 (1) — SAE. Abdominal pain following a study endoscopy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes